CLINICAL TRIAL: NCT05538858
Title: Vascular Injury in Mechanical Ventilation: a Proof-of-Concept Study
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Asher Mendelson, Assistant Professor, University of Manitoba
Other Study IDs: HS25427
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2023-05

CONDITIONS: Mechanical Ventilation Complication; Vascular Injury; Endothelial Dysfunction
MeSH Terms: conditions — Vascular System Injuries | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mechanical Ventilation: Cohort will undergo standard of care treatment utilizing a general anesthetic with mechanical ventilation for a surgical procedure.
  Interventions: Procedure: Mechanical Ventilation
- Control: Cohort will undergo standard of care treatment utilizing a regional or neuraxial anesthetic without mechanical ventilation for a surgical procedure.

INTERVENTIONS:
Procedure: Mechanical Ventilation — Positive pressure mechanical ventilation
  Groups: Mechanical Ventilation

SUMMARY:
Investigation of the effect of mechanical ventilation on biomarkers of microvascular damage

DETAILED DESCRIPTION:
The objective of this study is to determine the effect of mechanical ventilation (MV) on endothelial biomarkers associated with ventilator-induced vascular injury (VIVI), and determine the correlation of these biomarkers with non-invasive microvascular perfusion monitoring data and semaphorin 3E levels.

Blood samples will be collected immediately pre-operatively and post-operatively.

Biomarkers will be expressed as an absolute value and as a relative percentage change from baseline to account for inter-individual variability. Hemodynamic and surgical variables will be extracted from the OR data: blood pressure, oxygen saturation, blood loss, fluid administration, length of surgery, and MV parameters such as tidal volume, inspired oxygen, respiratory rate, and positive end-expiratory pressure.

During surgery, patients will be monitored using a non-invasive near-infrared spectroscopy technique to quantify skeletal muscle microvascular perfusion. These devices will be applied immediately prior to induction of anesthetic and data collected until immediately prior to transfer to the post-anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Patients undergoing elective orthopedic, endourologic, or plastic surgery procedure which is amenable to both general anesthetic or regional/neuraxial anesthesia

Exclusion Criteria:

* Emergency surgery
* Polytrauma
* Tourniquet use
* Controlled hypotension
* Mechanical ventilation less than 60 minutes in duration
* American Society of Anesthesiologists class 4 or greater
* Status postpneumonectomy
* Pulmonary hypertension
* Oxygen therapy during last month
* Severe obesity (body mass index ≥40 kg/m2)
* Immunosuppression within 3 months
* Diagnosed infection
* Shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective orthopedic, endourologic, or plastic surgery procedure amenable to both general anesthetic or regional/neuraxial anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Relative change of postoperative Granulocyte-macrophage colony-stimulating factor (GM-CSF) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interferon gamma (IFNγ) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-1β plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-1RA plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-2 plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-4 plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-5 plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-6 plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-8 plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-10 plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-12(p40) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-12(p70) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Interleukin-13 plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Monocyte Chemoattractant Protein-1 (MCP-1) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Tumor Necrosis Factor Alpha (TNFα) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Soluble platelet endothelial cell adhesion molecule-1 (sPECAM-1) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Vascular Cell Adhesion Molecule 1 (VCAM-1) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Vascular Endothelial Growth Factor (VEGF) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Angiopoietin 2 (Ang-2) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Tyrosine-protein kinase receptor Tie-2 (sTIE-2) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Soluble platelet selectin (sP-selectin) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Soluble endothelial selectin (sE-selectin) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative Soluble intercellular adhesion molecule-1 (sICAM-1) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative thrombomodulin plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure
Relative change of postoperative von Willebrand factor (vWF) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure

SECONDARY OUTCOMES:
Relative change of postoperative Semaphorin 3E (sema3E) plasma concentration relative to preoperative plasma concentration | Immediately prior to surgical procedure to immediately after surgical procedure
  Percentage change in concentration from immediately prior to surgical procedure to immediately after surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Asher Mendelson, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Center, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No